CLINICAL TRIAL: NCT01690468
Title: A Phase IA/IB Trial of PTX-200 and Carboplatin in Patients With Platinum-Resistant Recurrent Ovarian Cancer
Brief Title: PTX-200 and Carboplatin in Ovarian Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrollment stopped prior to Phase 1b, change in strategic focus
Sponsor: Prescient Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18641
Record Dates: First submitted 2012-09-19; First posted 2012-09-21 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — triciribine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triciribine & Carboplatin (Experimental): Phase I/II: 25mg/m^2 Triciribine and Carboplatin AUC 4. Triciribine escalated to 30, 35, 45mg/m^2 if toxicities are not encountered.
  Phase II: Recommended phase II dose of triciribine and carboplatin.
  Interventions: Drug: Triciribine; Drug: Carboplatin

INTERVENTIONS:
Drug: Triciribine — Triciribine (15, 25, 30, 35, or 45 mg/m^2) on days 1, 8, 15 every 21 days. To be given as a 60 minute IV infusion.
  Other Names: triciribine phosphate monohydrate; TCN; TCN-PM; AKT inhibitor
Drug: Carboplatin — Carboplatin will be administered on day 1 every 21 days, as a 30 minute IV infusion after completion of TCN.
  Other Names: Paraplatin®; NSC #241240

SUMMARY:
The main purpose of this study is to determine if Triciribine (TCN) and carboplatin are safe and tolerable when given together, and to determine if this combination of drugs can help people with recurrent ovarian cancer.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the safety and tolerability, and determine the maximum tolerated dose of triciribine when combined with carboplatin in women with platinum-resistant, recurrent or persistent ovarian cancer. The secondary objectives are to evaluate the clinical activity of carboplatin plus triciribine in women with recurrent/persistent, platinum-resistant ovarian cancer by assessing response rate, progression-free survival, and duration of stable disease.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Histologically confirmed, measurable or non-measurable, recurrent or persistent, platinum-resistant epithelial ovarian, fallopian tube or primary peritoneal carcinoma. By standard Gynecologic Oncology Group (GOG) criteria, platinum-resistant disease is defined by a disease-free interval of less than 6 months following treatment with a platinum-based regimen, or the progression of disease during platinum-based therapy.
* At least one prior regimen of chemotherapy, with no maximum number of chemotherapy cycles
* A serum creatinine ≤ 1.5 mg% obtained ≤ 2 weeks prior to entry
* Adequate hematologic reserve obtained ≤ 2 weeks prior to entry: leukocytes ≥ 3,000 mm^3; absolute neutrophil count ≥ 1500 mm^3; platelets ≥ 100,000 mm^3
* Adequate hepatocellular function: aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤ 3x upper limit of normal within institutional limits; bilirubin ≤ 1.5 mg/dl
* Gynecologic Oncology Group (GOG) Performance Status of 0, 1, or 2
* Life expectancy of at least 90 days
* The patient should be off chemotherapy, biologic therapy and radiation for 28 days.
* Neuropathy (sensory and motor) less than or equal to grade 1 per Common Toxicity Criteria (CTC) version 4

Exclusion Criteria:

* Prior TCN-PM therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to TCN-PM
* Patients must be disease-free of prior invasive malignancies for >2 years with the exception of basal cell or squamous cell carcinoma of the skin.
* Inability to give informed consent
* Pregnancy
* Corrected QT interval (QTc) prolongation > 450 milliseconds (msec)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 6 months
  To determine the maximum tolerated dose of TCN-PM when combined with carboplatin in a Phase I clinical trial of biomarker-selected women with platinum-resistant, recurrent or persistent epithelial ovarian, fallopian tube and primary peritoneal cancer (OVCA).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 2 years
  The best overall response is the best time point response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest sum recorded since baseline).
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm.
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Response and progression will be evaluated using Response Evaluation Criteria in Solid Tumors (RECIST version 1-1). Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.
Progression Free Survival (PFS) | 2 years
  Progression-Free Survival (PFS) is defined as the duration of time from study entry to time of progression or death, whichever occurs first.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
  Response and progression will be evaluated using Response Evaluation Criteria in Solid Tumors (RECIST version 1-1). Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.
Duration of Stable Disease (SD) | 2 years
  Stable Disease (SD): Neither sufficient shrinkage to qualify for Partial Response (PR) nor sufficient increase to qualify for Progressive Disease (PD), taking as reference the smallest sum diameters while on study.
  Response and progression will be evaluated using Response Evaluation Criteria in Solid Tumors (RECIST version 1-1). Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wenham, MD, Principal Investigator — H. Lee Moffitt Cancer Center
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No